CLINICAL TRIAL: NCT02210598
Title: Outpatient Labor Induction With the Transcervical Foley Balloon: A Randomized Trial Comparing Outpatient Immediate Removal Foley Versus Standard Inpatient Foley Induction
Brief Title: Outpatient Labor Induction With the Transcervical Foley Balloon
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Patrick M Mullin, MD, Associate Professor, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HS-13-00740
Record Dates: First submitted 2014-03-19; First posted 2014-08-06 (Estimated); Last update posted 2017-04-19 (Actual); Status verified 2017-04

CONDITIONS: Pregnancy; Labor; Forced or Induced, Affecting Fetus or Newborn
Keywords: labor, induced; catheter; oxytocin; Cesarean section
MeSH Terms: interventions — Oxytocin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- inpatient Foley balloon induction (Active Comparator): Inpatient Foley induction participants will be placed in the dorsal lithotomy position, a Foley catheter will be placed transcervically and its balloon filled with 60mL of sterile saline. One of two methods will be used to place the transcervical foley based on provider preference and determination of which method will offer the greatest chance for successful placement. Method A is placement of the foley "blindly" by palpation of the cervix. Method B utilizes direct visualization with sterile speculum placement. Method will be documented in the data collection forms. The catheter will be left in place and IV oxytocin will be started per LAC+USC protocol. The foley catheter will be removed after 12 hours if not spontaneously extruded.
  Interventions: Device: inpatient Foley balloon induction; Drug: Oxytocin
- outpatient Foley balloon induction (Experimental): Patients randomized to the experimental group will undergo outpatient Foley induction of labor. Either of the above two described methods will be used to place an 18 French Foley catheter transcervically and its balloon filled with 60mL of sterile saline. The catheter will be deflated and removed within 10 minutes of placement. The patient will then undergo a non-stress test (NST). If the patient has a reactive NST with no late or variable decelerations or uterine tachysystole, the patient will be discharged home with clear return precautions and instructions to return to the triage area in 24 hours. When the patient returns to the hospital, a sterile vaginal exam will be done and Bishop score documented. The patient will then be admitted to L&D for inpatient continuation of induction with IV oxytocin per LAC+USC protocol.
  Interventions: Device: outpatient Foley balloon induction; Drug: Oxytocin

INTERVENTIONS:
Device: inpatient Foley balloon induction — The catheter will be left in place and IV oxytocin will be started per LAC+USC protocol. The foley catheter will be removed after 12 hours if not spontaneously extruded.
  Other Names: 18-French Bard catheter
  Arms: inpatient Foley balloon induction
Device: outpatient Foley balloon induction — The catheter will be deflated and removed within 10 minutes of placement. The patient will then undergo a non-stress test (NST). If the patient has a reactive NST with no late or variable decelerations or uterine tachysystole, the patient will be discharged home with clear return precautions and instructions to return to the triage area in 24 hours.
  Other Names: 18-French Bard catheter
  Arms: outpatient Foley balloon induction
Drug: Oxytocin — When a patient randomized to the outpatient Foley Balloon induction group returns to the hospital, a sterile vaginal exam will be done and Bishop score documented. The patient will then be admitted to L&D for inpatient continuation of induction with IV oxytocin per LAC+USC protocol.
  Patients randomized to the inpatient Foley balloon induction group will have IV oxytocin initiated per LAC+USC protocol at the time of Foley balloon placement.

SUMMARY:
This study represents the first randomized trial comparing traditional inpatient induction with a transcervical foley catheter versus outpatient induction with immediate removal of a transcervical foley catheter. The immediate removal technique allows the induction process to begin in the hospital setting, but allows the patient to go home without a foreign body in situ. The investigators hypothesize the outpatient group will spend less time hospitalized prior to discharge. Additionally, the investigators will explore the vaginal delivery rates and maternal/neonatal safety profiles between groups.

DETAILED DESCRIPTION:
This is a randomized controlled trial.

Patients who are candidates for labor induction and meet inclusion criteria will be identified in the obstetrics clinic when they are being scheduled for induction of labor, or at a later clinic date. If they agree to participate, patients will be randomized and enrolled in the study at that time. Those who consent will be randomized into Group A (Experimental Group) and Group B (Control Group). No stratification criteria will be used.

Patients randomized to the control group will undergo induction of labor using the standard foley bulb and Pitocin method. Participants will be placed in the dorsal lithotomy position, an 18 French Foley catheter will be placed transcervically and its balloon filled with 60mL of sterile saline. One of two methods will be used to place the transcervical foley based on provider preference and determination of which method will offer the greatest chance for successful placement. Method A is placement of the foley "blindly" by palpation of the cervix. Method B utilizes direct visualization with sterile speculum placement. Method will be documented in the data collection forms. The catheter will be left in place and IV oxytocin will be started per protocol. The foley catheter will be removed after 12 hours if not spontaneously extruded.

Patients randomized to the experimental group will undergo outpatient induction of labor. Either of the above two described methods will be used to place an 18 French Foley catheter transcervically and its balloon filled with 60mL of sterile saline. The catheter will be deflated and removed within 10 minutes of placement. The patient will then undergo a non-stress test (NST). If the patient has a reactive NST with no late or variable decelerations or uterine tachysystole, the patient will be discharged home with clear return precautions and instructions to return to the triage area in 24 hours. When the patient returns to the hospital, a sterile vaginal exam will be done and Bishop score documented. The patient will then be admitted to L&D for inpatient continuation of induction with IV oxytocin per protocol.

In accordance with the Friedman curve and current LAC+USC practice, primigravid participants will be given 20 hours of maximum Pitocin (22 mU/ min) to achieve active labor and multigravid participants will be given 14 hours before a failed induction is diagnosed. Cesarean delivery will be recommended for arrest of dilation, arrest of descent, or any obstetric indication as decided by the on-duty house staff. Finally, at patient request, intravenous or regional anesthesia will be made available at any time during the labor and delivery process.

ELIGIBILITY:
Inclusion Criteria:

* Viable Intrauterine Pregnancy
* Greater than or equal to 37 weeks gestation on date of induction
* Cephalic Presentation
* Medically indicated induction of labor
* AFI greater than or equal to 5
* Patient able to be contacted by phone and demonstrates an understanding of the return instructions
* Cervical Dilation 2cm or less

Exclusion Criteria:

* Placenta Previa/Low Lying Placenta
* Placenta accreta/increta/percreta
* Undiagnosed vaginal bleeding
* Preeclampsia or HELLP Syndrome
* Intrauterine Growth Restriction
* Rupture of Membranes
* Prior cesarean section or transfundal uterine surgery
* Twin Gestation
* Fetal Anomaly
* Rh Isoimmunization
* Fetal Demise
* Uterine Tachysystole
* Less than 18 years of age
* HIV Infection
* Active herpes, hepatitis B or C infection
* Latex Allergy
* EFW>4000g
* Chorioamnionitis
* Non-English or Non-Spanish Speaking

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2014-03; Primary Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Duration of inpatient hospitalization (hours) | time from hospital admission to time to discharge, on average 96 hours
  compare inpatient time as measured by time from admission to time to discharge between the control (standard transcervical foley balloon placement/inpatient procedure) and the experimental group (immediate removal transcervical foley balloon placement/outpatient procedure)

SECONDARY OUTCOMES:
Duration of labor induction (hours) | time of initiation of labor induction to delivery, on average 24 hours
Cesarean section rate (percentage) | determined at time of delivery
Duration of oxytocin use during labor induction (hours) | time of initiation of oxytocin until it is discontinued, on average 18 hours
Rate of patients having prolonged fetal heart rate decelerations during labor induction (percentage) | from initiation of labor induction to delivery, on average 24 hours
Rate of patients developing chorioamnionitis during labor induction (percentage) | from initiation of induction until delivery, on average 24 hours
Rate of patients developing uterine tachysystole during labor induction (percentage) | from initiation of labor induction to delivery, on average 24 hours
Rate of infants admitted to NICU (percentage) | on average during the 24 hours following delivery
APGAR score | at 1 minute, 5 minutes, and 10 minutes after delivery

CONTACTS AND LOCATIONS:
Overall Officials: Patrick M Mullin, MD, Study Director — University of Southern California; Yen Chan, MD, Principal Investigator — University of Southern California; Richard Lee, MD, Study Director — University of Southern California
Locations (1):
- Los Angeles County + University of Southern California Medical Center, Los Angeles, California, United States

REFERENCES:
- [Result] Sciscione AC, Muench M, Pollock M, Jenkins TM, Tildon-Burton J, Colmorgen GH. Transcervical Foley catheter for preinduction cervical ripening in an outpatient versus inpatient setting. Obstet Gynecol. 2001 Nov;98(5 Pt 1):751-6. doi: 10.1016/s0029-7844(01)01579-4. PMID 11704164
- [Result] Kelly AJ, Alfirevic Z, Dowswell T. Outpatient versus inpatient induction of labour for improving birth outcomes. Cochrane Database Syst Rev. 2009 Apr 15;(2):CD007372. doi: 10.1002/14651858.CD007372.pub2. PMID 19370687
- [Result] Henry A, Madan A, Reid R, Tracy SK, Austin K, Welsh A, Challis D. Outpatient Foley catheter versus inpatient prostaglandin E2 gel for induction of labour: a randomised trial. BMC Pregnancy Childbirth. 2013 Jan 29;13:25. doi: 10.1186/1471-2393-13-25. PMID 23356673
- [Derived] de Vaan MD, Ten Eikelder ML, Jozwiak M, Palmer KR, Davies-Tuck M, Bloemenkamp KW, Mol BWJ, Boulvain M. Mechanical methods for induction of labour. Cochrane Database Syst Rev. 2023 Mar 30;3(3):CD001233. doi: 10.1002/14651858.CD001233.pub4. PMID 36996264
- [Derived] Alfirevic Z, Gyte GM, Nogueira Pileggi V, Plachcinski R, Osoti AO, Finucane EM. Home versus inpatient induction of labour for improving birth outcomes. Cochrane Database Syst Rev. 2020 Aug 27;8(8):CD007372. doi: 10.1002/14651858.CD007372.pub4. PMID 32852803